CLINICAL TRIAL: NCT01427595
Title: Effect of Metformin on Sensitivity of the GnRH Pulse Generator to Suppression by Estradiol and Progesterone in Hyperandrogenemic Adolescent Girls (JCM025)
Brief Title: Effect of Metformin on Sensitivity of the GnRH Pulse Generator to Suppression by Estradiol and Progesterone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Christine Burt Solorzano, Center for Research in Reproduction, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13789; U54HD028934-18 (NIH)
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Results first posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-12

CONDITIONS: Polycystic Ovary Syndrome; Hyperandrogenism
Keywords: hyperandrogenemia
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperandrogenism | interventions — Metformin; Progesterone; Estradiol; Estrogens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin, progesterone , estrace (Experimental): 12 weeks Metformin oral progesterone suspension (20 mg/ml, 25-100 mg) three times a day at 0700, 1500, and 2300 hr for seven days (2X) oral estrace, 0.5-1 mg once a day for seven days (2X)
  Interventions: Drug: Metformin; Drug: Progesterone; Drug: estrace

INTERVENTIONS:
Drug: Metformin — 500-2000 mg PO BID (X12 weeks)
Drug: Progesterone — oral progesterone suspension (20 mg/ml, 25-100 mg) three times a day at 0700, 1500, and 2300 hr for seven days (X2)
Drug: estrace — oral estrogen (estrace, 0.5-1 mg once a day for seven days)- X2
  Other Names: Estrogen

SUMMARY:
Many, but not all, girls with high levels of the male hormone testosterone go on to develop polycystic ovary syndrome (PCOS) as adults. Women with PCOS often have irregular menstrual periods, excess facial and body hair, and weight gain. PCOS is also a leading cause of difficulty becoming pregnant. The investigators do not understand why some girls with high hormones develop PCOS and others do not. In a previous study by our group, some girls with high levels of male hormones had abnormalities in the secretion of another hormone, called luteinizing hormone (LH), that are often seen in women with PCOS. However, another group had normal LH secretion. The girls with the abnormal LH secretion had higher levels of another hormone, called insulin, than the girls with normal LH secretion. The investigators will test whether metformin, an insulin-sensitizing agent, changes the effects of high male hormone levels in adolescent girls, specifically by looking at their LH secretion response following metformin treatment.

DETAILED DESCRIPTION:
A better understanding of the factors that make adolescent girls more or less susceptible to the adverse neuroendocrine effects of elevated androgens will hopefully lead to improved prevention and treatment strategies for PCOS. In this study, we propose to explore the role of hyperinsulinemia on neuroendocrine function in hyperandrogenic adolescent girls by assessing the effect of the insulin sensitizer Metformin on hypothalamic progesterone sensitivity. Other differences between the progesterone sensitive and progesterone insensitive subgroups, including racial and ethnic differences between the two populations and a trend towards older gynecologic age in the progesterone insensitive population, are being pursued through other ongoing studies (IRB-HSR# 8588 and 12160).

ELIGIBILITY:
Inclusion Criteria:

* Girls ages 10 to 17
* Hyperandrogenemic (free testosterone greater than 2.5 standard deviations above the mean for normal control subjects of the same Tanner Stage)
* Creatinine clearance > 90 ml/min as calculated by the Cockcroft-Gault equation
* Hemoglobin > 12 mg/dL or Hematocrit > 36%
* Normal screening labs (with exception of the expected hormonal abnormalities inherent in hyperandrogenemia)
* Sexually active subjects must agree to abstain or use double barrier contraception during the study
* Subjects must agree not to take any other medications during the course of the study without approval by the study investigators.

Exclusion Criteria:

* Abnormal screening labs (with the exception of the expected hormonal abnormalities inherent in hyperandrogenemia)
* Creatinine clearance less than 90 ml/min as calculated by Cockcroft-Gault equation
* Hemoglobin <12 mg/dL or hematocrit < 36%
* Abnormal liver function tests, including Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Bilirubin, Albumin, and Alkaline Phosphatase
* Weight < 34 kg
* History of renal dysfunction, liver dysfunction, congestive heart failure, deep venous thrombosis, breast cancer, endometrial cancer, or cervical cancer
* Pregnant or breast feeding
* On medications known to affect the reproductive axis within 3 months of the study (including oral contraceptive pills, metformin, and spironolactone)
* Are currently participating in another study or have been in one in the last 30 days.
* Subjects using restricted medication (see restrictions below) are excluded unless the subject's primary care provider approves stopping the medication.

Ages: 10 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2009-02-18 (Actual); Primary Completion 2015-01-17 (Actual); Study Completion 2015-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C. Marshall, MD, PhD, Principal Investigator — University of Virginia
Locations (1):
- Center for Research in Reproduction, University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Lundgren JA, Kim SH, Burt Solorzano CM, McCartney CR, Marshall JC. Progesterone Suppression of Luteinizing Hormone Pulse Frequency in Adolescent Girls With Hyperandrogenism: Effects of Metformin. J Clin Endocrinol Metab. 2018 Jan 1;103(1):263-270. doi: 10.1210/jc.2017-02068. PMID 29095983

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 25 subjects enrolled in this study. 7 subjects completed screening procedures only (these 7 subjects were withdrawn from study prior to being assigned to an arm of intervention).
Period: Overall Study
Arm/Group | Metformin, Progesterone , Estrace
Started | 25
Completed | 12
Not Completed | 13

BASELINE CHARACTERISTICS:
Population: 25 subjects enrolled and 12 completed the study. Only 10 subjects were included in the formal analysis.
Arm/Group | Metformin, Progesterone , Estrace
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.3 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Progesterone Sensitivity Index Before and After Metformin Treatment.
Description: The progesterone (P4) sensitivity index is defined as the percent change in 11-hour LH pulse frequency before and after P4 and estradiol administration for 7 days, divided by the day 7 mean serum P4 concentration. We compared the P4 sensitivity index after metformin administration to the baseline P4 sensitivity index, using Wilcoxon signed-rank test.
Time Frame: 12 weeks following start of metformin treatment
Population: 12 subjects completed study but 2 subjects were excluded from analysis due to incomplete adherence to metformin, missing > 10% of doses.
Measure: Mean (Standard Deviation); unit: % change in LH pulses/day 7 P4 level
Arm/Group | Metformin, Progesterone , Estrace
Number analyzed (Participants) | 10
% change in LH pulses/day 7 P4 level
  Before Metformin | -4.12 (2.39)
  After Metformin | -4.29 (7.66)

ADVERSE EVENTS:
Time Frame: From start of study procedures until 30 days post study drug.
Arm/Group | Metformin, Progesterone , Estrace
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 12/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin, Progesterone , Estrace (N=25)
Vision switched from near to farsighted (Eye disorders) | 1 (1)
SVT (Cardiac disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
headache (General disorders) | 1 (1)
nausea (General disorders) | 2 (2)
UTI (Infections and infestations) | 3 (3)
fainting (General disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 2 (2)
Acute Gastroenteritis (Gastrointestinal disorders) | 1 (1)
heartburn (General disorders) | 1 (1)
vomitting (Gastrointestinal disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-12-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT01427595/Prot_SAP_000.pdf
  • Informed Consent Form (2015-12-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT01427595/ICF_001.pdf